CLINICAL TRIAL: NCT02239822
Title: Double Blinded Randomized Trial of eTNS as Adjuvant Treatment for Major Unipolar Depressive Disorder.
Brief Title: Electrical Stimulation in Patients With Unipolar Major Depression
Acronym: TREND2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 271/2013
Record Dates: First submitted 2014-08-21; First posted 2014-09-15 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Depression
Keywords: Electrodes, Implanted; Electric Stimulation Therapy
MeSH Terms: conditions — Depression | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Stimulation (Active Comparator): Patients assigned to active stimulation arm will receive electrical stimulation during the study.
  Interventions: Procedure: Stimulation of the trigeminal nerve (active stimulation)
- Placebo Stimulation (Placebo Comparator): Patients assigned to the placebo arm did not receive stimulation electrical stimulation for 24 weeks. After this period the participants randomized to sham stimulation will be moved to the active stimulation and will be followed until study completion.
  Interventions: Procedure: Placebo stimulation of the trigeminal nerve (placebo)

INTERVENTIONS:
Procedure: Stimulation of the trigeminal nerve (active stimulation) — Participants will be randomized to active vs. sham stimulation during a period of 24 weeks with a one-way cross over at 12 weeks.
  After 12 weeks, the participants receiving active electrical stimulation will continue under active stimulation until completion of the study.
  Participants randomized to sham stimulation will be shifted to active stimulation and will be followed-up until completion of the study.
  The study will be unblinded after 6 months of randomized stimulation. The second part of the study will be an open label prospective trial for evaluate long-term follow-up. The duration of the open label trial will be more 24 weeks. the duration of the open label trial will be more 24 weeks.
  Other Names: Electrical Stimulation
  Arms: Active Stimulation
Procedure: Placebo stimulation of the trigeminal nerve (placebo) — Participants will be randomized to active vs. sham stimulation during a period of 24 weeks with a one-way cross over at 12 weeks.
  After 12 weeks, the participants receiving active electrical stimulation will continue under active stimulation until completion of the study.
  Participants randomized to sham stimulation will be shifted to active stimulation and will be followed-up until completion of the study.
  The study will be unblinded after 6 months of randomized stimulation. The second part of the study will be an open label prospective trial for evaluate long-term follow-up. The duration of the open label trial will be more 24 weeks.
  Other Names: Sham Eletrical Stimulation
  Arms: Placebo Stimulation

SUMMARY:
Double Blinded Randomized Trial of eTNS as adjuvant treatment for Major Unipolar Depressive Disorder. The primary objective is to assess the safety and tolerability of eTNS (external trigeminal nerve stimulation) of the V1 branch of the trigeminal nerve as an adjunctive treatment for adult patients with the diagnosis of unipolar MDD (Major Depressive Disorder).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with non-psychotic, unipolar Major Depressive Disorder assessed via the MINI structured interview and legally capacitated to sign the informed consent for participation in the study;
* A score of ≥ 14 on the HAM-D17 with Item 1 (depressed mood) ≥ 2;
* A history of treatment failure with at least 3 adequate trials antidepressants over the previous 6 weeks and less than 6 medications, with no change in antidepressant medication or dose within the previous 6 weeks, and ongoing use of at least one antidepressant (which will continue during participation in the study);
* Patients with suicidal ideation are eligible only if the thoughts of death or of life not being worth living are not accompanied by a plan or intention for self-harm and lack of self-harming attempt in the past 6 months;
* Patients with appropriate support to be compliant with the study protocol.

Exclusion Criteria:

* Patient is mentally or legally incapacitated, unable to give informed consent;
* Patients with psychosis (psychotic depression, schizophrenia, or schizoaffective diagnoses (lifetime); bipolar disorder (lifetime); dementia (lifetime); delirium or any substance abuse disorder within the past 6 months; eating disorder within the past year; obsessive-compulsive disorder (lifetime); post-traumatic stress disorder within the past year; acute risk for suicide or self-injurious behavior. Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudo-dementia of depression) will be excluded;
* Patients currently receiving more than six medications for treatment of MDD;
* Patients with exposure to ECT or rTMS or any investigational treatment (for any disorder) within the past 6 months;
* Prior VNS and/or DBS therapy (lifetime);
* Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke, CVA, or TIAs; cerebral aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
* Current pregnancy, breast feeding, plans to become pregnant during the study, or not using a medically accepted means of contraception;
* Other medical conditions that would increase the risk of infection or surgical related morbidity and/or would affect compliance with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Identify a efficacy of eTNS of the V1 branch of the trigeminal nerve | 48 weeks
  We will use the Hamilton Rating Scale for Depression (HRSD) 17 scores as the main outcome measure to assess the efficacy of sTNS of the V1 branch of the trigeminal nerve as adjunctive treatment for MDD.

SECONDARY OUTCOMES:
Identify the tolerability of eTNS stimulation | 48 weeks
  Tolerability will be evaluated by the records of adverse effects observed during the randomized, open stimulation. We will apply the Ugvalg for Kliniske Undersgelser (UKU) scale at all visits for all patients and to compare scores between groups. Adverse events will be categorized using the MedDRA Medical Dictionary for Regulatory Activities. Complications reported by active and sham stimulation groups will be compared. The complication risk will be calculated based on the overall study duration.
Identify the long-term recurrence rate of eTNS therapy | 48 weeks
  We will calculate the recurrence rate of all participants at the end of the open label prospective follow-up. Recurrence is defined as return of HAM-17 scores equal to or superior to the original, after the patient has lodged during partial response (20% decrease of the initial score) or complete response (50% decrease of the initial score).
Identify the duration of the placebo effect | 48 weeks
  To evaluate the duration of the placebo effect in participants randomized to sham stimulation during the initial 12 weeks of the trial. The mean, median and the standard deviation of the interval time to recurrence will be calculated on placebo stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gorgulho, MD, MSc, Principal Investigator — HOSPITAL DO CORAÇÃO; Antonio De Salles, M.D., Ph.D., Principal Investigator — HOSPITAL DO CORAÇÃO; Otavio Berwanger, MD,PhD, Study Director — HOSPITAL DO CORAÇÃO
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil